CLINICAL TRIAL: NCT04014686
Title: Impacts of 12 Weeks of Resistance Band Exercise Training on Insulin Resistance, Blood Lipids, Body Composition, and Blood Pressure in Postmenopausal Women With Obesity
Brief Title: 12 Weeks of Resistance Band Exercise Impacts on Metabolic Syndrome Progression in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Dong-Eui University (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UNOmaha9
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Metabolic Syndrome; Dyslipidemias; Insulin Resistance; Hypertension
Keywords: postmenopausal; exercise
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias; Insulin Resistance; Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: exercise intervention group, control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): No exercise intervention
  Interventions: Other: No exercise intervention group
- Exercise intervention group (Experimental): Exercise intervention group (resistance band exercise training for 12 weeks, 3x per week, for 60 minutes per day).
  Interventions: Behavioral: Resistance band exercise intervention group

INTERVENTIONS:
Other: No exercise intervention group — no exercise intervention
  Arms: Control group
Behavioral: Resistance band exercise intervention group — Resistance band exercise training intervention (12 weeks, 3x per week, for 60 minutes per day)
  Arms: Exercise intervention group

SUMMARY:
The purpose of this study was to examine the impacts of a 12-week resistance band exercise program on insulin resistance, blood lipid profiles, body composition, and blood pressure in postmenopausal women with obesity.

Thirty-six postmenopausal women participated in this study. Participants were randomly allocated into the resistance band training group (EX, n = 18) or the control group (CON, n = 18). The EX group performed a resistance band exercise training program 60 minutes per day, 3 times per week, for 12 weeks. The CON group did not participate in any exercise, dietary, or behavioral intervention. Blood glucose, insulin, homeostatic model of insulin resistance (HOMA-IR), blood lipids, blood pressure, and body composition were measured before and after 12 weeks of EX or CON.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal (cessation of menses for at least 12 consecutive months)
* abdominal obesity (waist > 80 cm)

Exclusion Criteria:

* current smoker (smoking within 6 months of participation)
* cardiovascular disease
* renal disease
* pulmonary disease
* thyroid disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female, postmenopausal
Enrollment: 36 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Glucose | 12 weeks
  Blood glucose was measured before and after 12 weeks.
Insulin | 12 weeks
  Blood insulin was measured before and after 12 weeks.
Percentage of Body Fat | 12 weeks
  Body fat percentage was measured before and after 12 weeks.
Waist circumference | 12 weeks
  Waist circumference was measured before and after 12 weeks.

SECONDARY OUTCOMES:
Systolic blood pressure | 12 weeks
  Systolic blood pressure was measured before and after 12 weeks.
Diastolic blood pressure | 12 weeks
  Diastolic blood pressure was measured before and after 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No